CLINICAL TRIAL: NCT04602728
Title: Building Adaptive Coping and Knowledge to Improve Daily Life (Back2Life): A Pilot Feasibility Clinical Trial for Youth With Chronic Sickle Cell Pain
Brief Title: Building Adaptive Coping and Knowledge to Improve Daily Life
Acronym: Back2Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Soumitri Sil, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00000573; 1K23HL133457 (NIH); R03HL164333 (NIH)
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Sickle Cell Disease
Keywords: Pediatrics; Cognitive behavioral therapy; Behavioral intervention
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Youth and parent/caregiver dyads will participate in the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Back2Life Program (Experimental): Youth with chronic SCD pain and their parents or caregivers receiving an adaptive cognitive behavioral treatment program for pain coping skills.
  Interventions: Behavioral: Back2Life

INTERVENTIONS:
Behavioral: Back2Life — The Back2Life intervention uses an adaptive treatment approach with module-based treatment sessions selected on the basis of baseline assessment (rather than a fixed treatment approach) to allow flexibility in tailoring treatment components to meet individual family needs. All youth participants will receive the standard 6-session pain coping skills training program, consisting of learning ways to cope with and manage chronic sickle cell pain. The standard program includes topics that were identified by young people with chronic sickle cell pain and their parents as important skills for all youth with chronic pain and sickle cell disease. In addition to the standard 6-session program, youth participants may receive an additional 1 to 4 sessions that may help with specific problems and/or co-morbidities related to pain. At least one parent or guardian is required to attend the sessions with their child.

SUMMARY:
The purpose of this study is to find out how teenagers with chronic pain and sickle cell disease respond to a new training program called Back2Life and get their feedback about how to modify the program to best fit their needs. The Back2Life training program focuses on teaching pain coping skills (also known as cognitive-behavioral therapy). The program teaches skills and strategies that may help teens improve chronic pain management and get back into their everyday activities.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is a genetic disorder of the hemoglobin in which the course of acute pain from vaso-occlusion and its sequelae vary widely across genotypes and individual patients. SCD pain often begins during childhood and can progress to chronic pain for approximately 23% of children and adolescents. Youth with chronic SCD pain, that is pain that is present on most days per month and persists for at least 6 months, report high levels of functional disability, elevated depressive and anxiety symptoms, and reduced quality of life relative to youth with SCD without chronic pain. The complex, multifactorial nature of chronic SCD pain can also contribute to increased healthcare utilization for pain. The most effective management and treatment of chronic SCD pain likely requires individualized, multimodal, multidisciplinary treatments that go beyond pharmacological management alone. A range of evidence-based non-pharmacological treatments, such as behavioral health, complementary, and integrative health approaches, are recommended for chronic pain management and are gaining greater awareness and integration into comprehensive chronic pain care.

Behavioral health treatment, such as cognitive-behavioral therapy (CBT) for pain, focuses on improved daily functioning and coping through several core treatment components such as psychoeducation about how the body processes pain, relaxation skills training, and cognitive strategies. Youth with chronic SCD pain need an evidence-based, culturally informed, adaptive treatment. Behavioral treatments that are tailored to patient and family needs are beneficial when patients may require different levels of care. Adaptive designs are more effective in improving health outcomes, satisfaction with treatment, and reducing healthcare use than standard protocols where patients receive a fixed "one size fits all" treatment that is not personalized to their needs; adaptive designs are also recommended for tailoring evidence-based interventions with culturally diverse populations. Adaptive treatments can integrate evidence-based strategies to address common co-morbid problems associated with chronic pain, such as elevated anxiety or depressive symptoms or sleep disturbance. Teaching parents problem-solving skills can reduce caregiver stress among families managing chronic pain and illness.

This study utilizes an adaptive behavioral treatment to target psychosocial risk factors for youth with chronic SCD pain as a first step towards developing a stepped care model for SCD pain. The proposed treatment, called Back2Life, is innovative because it is culturally informed by families' and patients' feedback regarding their treatment preferences and targets psychological co-morbidities that are often excluded in clinical trials. The overarching hypothesis driving the proposed intervention is that disrupting the complex interacting psychosocial factors that can exacerbate chronic SCD pain will prevent and/or reduce poor health outcomes in children and adolescents with SCD. Reductions in inflammatory biomarkers are examined as an exploratory hypothesis and participants can consent to an optional blood draw for this portion of the study.

ELIGIBILITY:
Inclusion Criteria for Youth:

* diagnosed with SCD (any genotype)
* report chronic pain
* speak and read English
* have not initiated new disease modifying-treatments (e.g, hydroxyurea, Endari, voxelotor, crizanlizumab, chronic transfusions) or significantly increased dosages of any disease-modifying treatments in the past 3 months

Inclusion Criteria for Parents or Caregivers:

* speak and read English

Exclusion Criteria for Youth:

* have comorbid medical conditions typically associated with pain but unrelated to SCD (e.g., rheumatologic disorders or inflammatory bowel disease)
* are receiving chronic transfusion indicated for central nervous system risks and/or complications, previous overt strokes, or significant cognitive or developmental limitations, as per their healthcare provider or parent, that would impair completion of self-report measures or engagement in treatment sessions
* received ≥ 3 sessions of outpatient psychological therapy for pain management in the 6 months prior to screening

Exclusion Criteria for Parents or Caregivers:

* have significant cognitive limitations or severe psychiatric conditions, as per the child's healthcare team or history, that would impair completion of self-report measures or engagement in treatment sessions

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2024-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soumitri Sil, PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Children's Healthcare of Atlanta at Hughes Spalding, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory Children's Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Children's Healthcare of Atlanta, Emory Children's Center, and Children's Healthcare of Atlanta at Hughes Spalding in Atlanta, Georgia, USA. Participant enrollment began January 27, 2021. Data collection for the 6 Month time point ended August 23, 2023 and data collection for the 12 Month time point was complete on May 18, 2024.
Groups:
- Back2Life Program for Youth: Youth with chronic sickle cell disease (SCD) pain receiving an adaptive cognitive behavioral treatment program for pain coping skills.
- Back2Life for Parents or Caregivers: Parents or caregivers of youth with chronic SCD pain receiving an adaptive cognitive behavioral treatment program for pain coping skills.
Period: Overall Study
Arm/Group | Back2Life Program for Youth | Back2Life for Parents or Caregivers
Started | 20 | 20
Completed the Study Treatment of the Entire Back2Life Program | 16 | 16
Completed | 16 | 16
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Back2Life Program for Youth: Youth with chronic SCD pain receiving an adaptive cognitive behavioral treatment program for pain coping skills.
- Total: Total of all reporting groups
Arm/Group | Back2Life Program for Youth | Back2Life for Parents or Caregivers | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.8 (1.7) | 41.6 (5.1) | 26.9 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 19 | 28
  Male | 11 | 1 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 15 | 33
  Unknown or Not Reported | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 15 | 35
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 5 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) Pediatric Short Form Pain Interference Score
Description: The PROMIS Pediatric Short Form for Pain Interference, Self- and Parent-Proxy Report, is an 8-item self-report measure assessing functional interference due to pain in the past 7 days. Total scores are standardized to a T-score with a mean of 50 and a standard deviation of 10, where higher scores indicate increased hindrance of life activities due to pain.
Time Frame: Baseline, Immediately Post-Treatment, Month 3, Month 6
Population: The analysis population includes participants remaining in the study at the indicated time points.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Back2Life Program for Youth | Back2Life for Parents or Caregivers
Number analyzed (Participants) | 20 | 20
T-score
  Baseline | 61.5 (10.8) | 62.1 (11.1)
  Immediately Post-Treatment: number analyzed (Participants) | 16 | 16
  Immediately Post-Treatment | 58.2 (12.5) | 59.4 (12.2)
  Month 3: number analyzed (Participants) | 16 | 16
  Month 3 | 50.4 (11.6) | 53.7 (12.9)
  Month 6: number analyzed (Participants) | 16 | 16
  Month 6 | 50.3 (14.1) | 57.7 (11.9)

2. Primary Outcome: Sickle Cell Disease Pain Burden Interview-Youth (SCPBI-Y) Score
Description: The Sickle Cell Pain Burden Interview for Youth, Self-Report is a 7-item, validated measure of pain burden in 7-21 year olds. Responses are given on a 5-point Likert scale where 0 = none and 4 = every. The patient self-reports the amount of days in the past month where pain occurred or pain impacted daily life. Total scores range from 0 to 28 and higher scores indicate a greater pain burden.
Time Frame: Baseline, Immediately Post-Treatment, Month 3, Month 6
Population: The analysis population includes youth participants remaining in the study at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Back2Life Program for Youth
Number analyzed (Participants) | 20
score on a scale
  Baseline | 13.8 (7.5)
  Immediately Post-Treatment: number analyzed (Participants) | 16
  Immediately Post-Treatment | 9.5 (7.7)
  Month 3: number analyzed (Participants) | 16
  Month 3 | 9.1 (5.3)
  Month 6: number analyzed (Participants) | 16
  Month 6 | 7.0 (7.0)

3. Primary Outcome: PROMIS Pediatric Short Form Pain Behaviors, Parent-Proxy Report Score
Description: The PROMIS Pediatric Short Form Pain Behaviors, Parent-Proxy Report is an 8-item measure completed by parents that assesses pain behaviors displayed by their child in the past 7 days. Total scores are standardized to a T-score with a mean of 50 and a standard deviation of 10, where higher scores indicate increased behaviors due to pain.
Time Frame: Baseline, Immediately Post-Treatment, Month 3, Month 6
Population: The analysis population includes parent or caregiver participants remaining in the study at the indicated time points.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Back2Life for Parents or Caregivers
Number analyzed (Participants) | 20
T-score
  Baseline | 52.7 (20.6)
  Immediately Post-Treatment: number analyzed (Participants) | 16
  Immediately Post-Treatment | 52.0 (20.6)
  Month 3: number analyzed (Participants) | 16
  Month 3 | 46.2 (22.0)
  Month 6: number analyzed (Participants) | 16
  Month 6 | 50.8 (25.9)

4. Primary Outcome: Child Self-Efficacy Scale Score
Description: Child Self-Efficacy Scale, Self- and Parent-Proxy Report is a well-established, 7-item measure of self-efficacy for functioning despite pain for 8-19 year olds. Respondents report how sure about their (or their child's) ability to perform certain daily tasks when they have pain, on a scale from 1 to 5 where 1 = very sure and 5 = very unsure. Total scores range from 7 to 35 and lower scores indicate greater self-efficacy.
Time Frame: Baseline, Immediately Post-Treatment, Month 3, Month 6
Population: The analysis population includes participants remaining in the study at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Back2Life Program for Youth | Back2Life for Parents or Caregivers
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 23.0 (8.5) | 24.6 (8.2)
  Immediately Post-Treatment: number analyzed (Participants) | 16 | 16
  Immediately Post-Treatment | 20.0 (5.8) | 24.1 (8.1)
  Month 3: number analyzed (Participants) | 16 | 16
  Month 3 | 18.3 (2.6) | 24.3 (5.5)
  Month 6: number analyzed (Participants) | 16 | 16
  Month 6 | 17.0 (4.0) | 21.6 (8.9)

5. Primary Outcome: Number of Dyads Completing the Study
Description: Treatment feasibility was assessed by the number of participant dyads who complete the study.
Time Frame: Month 6
Measure: Count of Units; unit: dyads
Units Other Than Participants: dyads
Groups:
- Back2Life for Youth and Caregiver Dyads: Youth with chronic SCD pain and their parents or caregivers who are receiving an adaptive cognitive behavioral treatment program for pain coping skills.
Arm/Group | Back2Life for Youth and Caregiver Dyads
Number analyzed (Participants) | 40
Number analyzed (dyads) | 20
dyads | 16

6. Primary Outcome: Number of Dyads Completing Study Assignments Within Six Months
Description: Treatment feasibility was assessed by the number of dyads completing the 6-Month study assignment.
Time Frame: Month 6
Population: The analysis population includes youth and caregivers dyad participants who completed the Back2Life program.
Measure: Count of Units; unit: dyads
Units Other Than Participants: dyads
Groups:
- Back2Life for Youth and Caregiver Dyads: Youth with chronic SCD pain, and their parents or caregivers, who are receiving an adaptive cognitive behavioral treatment program for pain coping skills.
Arm/Group | Back2Life for Youth and Caregiver Dyads
Number analyzed (Participants) | 40
Number analyzed (dyads) | 20
dyads | 16

7. Primary Outcome: Number of Participants With Positive Experiences During Participant Evaluation of the Intervention Interview
Description: Treatment feasibility was assessed via a qualitative interview where participants were asked open ended questions. Participants were asked if they thought the Back2Life program helpful, if delivering the program through telemedicine was reasonable, and if the program was a reasonable approach for chronic pain management of sickle cell disease.
Time Frame: Immediately Post-Treatment
Population: The analysis population includes participants who completed the Back2Life program.
Measure: Count of Participants; unit: Participants
Arm/Group | Back2Life Program for Youth | Back2Life for Parents or Caregivers
Number analyzed (Participants) | 16 | 16
Participants
  Reported program was helpful | 15 | 16
  Reported a positive experience with telehealth delivery | 16 | 16
  Reported the program was relevant to sickle cell disease | 16 | 16

8. Primary Outcome: Treatment Evaluation Inventory-Short Form (TEI-SF) Score
Description: The Treatment Evaluation Inventory-Short Form was completed at the end of treatment. It includes 9 items adapted to be specific to pediatric pain. Items are rated on a 5-point Likert scale ranging from 1 to 5. Total scores range from 9 to 45. Higher scores indicate increased acceptability with the study treatment.
Time Frame: Immediately Post-Treatment
Population: The analysis population includes participants who completed the Back2Life program.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Back2Life Program for Youth | Back2Life for Parents or Caregivers
Number analyzed (Participants) | 16 | 16
score on a scale | 32.0 (6.1) | 31.5 (4.3)

9. Secondary Outcome: Emergency Department Visits Per Participant
Description: Healthcare utilization was extracted from the medical record to document the mean number of emergency department (ED) visits for pain per participant during the 12 months preceding the intervention period and the 12-month period post-treatment.
Time Frame: 12 months prior to Baseline, 12 months post-treatment
Measure: Mean (Standard Deviation); unit: visits per participant
Arm/Group | Back2Life Program for Youth
Number analyzed (Participants) | 20
visits per participant
  12 Months Pre-Treatment | 0.86 (1.06)
  12 Months Post-Treatment | 0.9 (1.07)

10. Secondary Outcome: Hospital Admissions Per Participant
Description: Healthcare utilization was extracted from the medical record to document the mean number of hospital admissions for pain per participant during the 12 months preceding the intervention and the 12-month period post-treatment.
Time Frame: 12 months prior to Baseline, 12 months post-treatment
Measure: Mean (Standard Deviation); unit: admissions per participant
Arm/Group | Back2Life Program for Youth
Number analyzed (Participants) | 20
admissions per participant
  12 Months Pre-Treatment | 1.19 (1.29)
  12 Months Post-Treatment | 1.25 (1.29)

11. Secondary Outcome: Days Per Week of Opioid Use
Description: Daily use of opioid pain medication was determined based on participant completion of daily diaries for 1-week at each assessment visit. Participants recorded opioid use daily (presence/absence).
Time Frame: Baseline, Immediately Post-Treatment, Month 3, Month 6
Population: The analysis population includes youth participants remaining in the study at the indicated time points.
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Back2Life Program for Youth
Number analyzed (Participants) | 20
days/week
  Baseline | 3.9 (2.1)
  Immediately Post-Treatment: number analyzed (Participants) | 16
  Immediately Post-Treatment | 1.5 (1.4)
  Month 3: number analyzed (Participants) | 16
  Month 3 | 1.8 (0.75)
  Month 6: number analyzed (Participants) | 16
  Month 6 | 1.2 (0.75)

12. Secondary Outcome: Pediatric Inventory for Parents (PIP) Score
Description: The Pediatric Inventory for Parents is a 42-item parent-reported measure of caregiver stress related to child chronic illness. Responses are given on a 5-point Likert scale where 1 = not at all and 5 = extremely. Total scores range from 42 to 210 and higher scores indicate greater caregiver stress.
Time Frame: Baseline, Immediately Post-Treatment, Month 3, Month 6
Population: The analysis population includes participants remaining in the study at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Back2Life for Parents or Caregivers
Number analyzed (Participants) | 20
score on a scale
  Baseline | 104.5 (29.3)
  Immediately Post-Treatment: number analyzed (Participants) | 16
  Immediately Post-Treatment | 91.0 (46.7)
  Month 3: number analyzed (Participants) | 16
  Month 3 | 72.0 (39.8)
  Month 6: number analyzed (Participants) | 16
  Month 6 | 71.0 (32.0)

13. Secondary Outcome: Adolescent Sleep Wake Scale (ASWS) Score
Description: The Adolescent Sleep Wake Scale (ASWS) is a 28-item patient-reported describing the occurrence and frequency of various behavioral sleep characteristics over the past month. Responses are given on a 6-point Likert scale where 1 = always and 6 = never. Total scores are calculated as the mean score from each time and range from 1 to 6 where higher scores indicate better sleep quality.
Time Frame: Baseline, Immediately Post-Treatment, Month 3, Month 6
Population: The analysis population includes participants remaining in the study at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Back2Life Program for Youth
Number analyzed (Participants) | 20
score on a scale
  Baseline | 2.9 (0.4)
  Immediately Post-Treatment: number analyzed (Participants) | 16
  Immediately Post-Treatment | 3.1 (0.5)
  Month 3: number analyzed (Participants) | 16
  Month 3 | 2.8 (0.2)
  Month 6: number analyzed (Participants) | 16
  Month 6 | 3.0 (0.3)

14. Secondary Outcome: PROMIS Pediatric Short Form Depressive Symptoms Score
Description: The PROMIS Pediatric Short Form Depressive Symptoms questionnaire, Self- and Parent-Proxy Report is an 8-item measure designed for youth to assess self-reported symptoms of depression. Total scores are standardized to a T-score with a mean of 50 and a standard deviation of 10, where higher scores indicate increased depression.
Time Frame: Baseline, Immediately Post-Treatment, Month 3, Month 6
Population: The analysis population includes participants remaining in the study at the indicated time points.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Back2Life Program for Youth | Back2Life for Parents or Caregivers
Number analyzed (Participants) | 20 | 20
T-score
  Baseline | 71.1 (6.3) | 55.4 (10.9)
  Immediately Post-Treatment: number analyzed (Participants) | 16 | 16
  Immediately Post-Treatment | 68.9 (7.0) | 52.6 (16.2)
  Month 3: number analyzed (Participants) | 16 | 16
  Month 3 | 65.5 (4.9) | 48.2 (12.0)
  Month 6: number analyzed (Participants) | 16 | 16
  Month 6 | 65.1 (4.5) | 47.9 (12.3)

15. Secondary Outcome: Pain Catastrophizing Scale Score
Description: The Pain Catastrophizing Scale, Child and Parent Report, is a 13-item well-validated self-report and parent-report measure of worried thoughts about pain. Items are answered on a 5-point scale where 0 = not true at all and 4 = very true. Total scores range from 0 to 52 and higher scores indicate increased catastrophic thinking.
Time Frame: Baseline, Immediately Post-Treatment, Month 3, Month 6
Population: The analysis population includes participants remaining in the study at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Back2Life Program for Youth | Back2Life for Parents or Caregivers
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 27.8 (12.0) | 33.3 (12.4)
  Immediately Post-Treatment: number analyzed (Participants) | 16 | 16
  Immediately Post-Treatment | 24.9 (10.7) | 35.8 (15.3)
  Month 3: number analyzed (Participants) | 16 | 16
  Month 3 | 18.1 (7.2) | 25.6 (13.7)
  Month 6: number analyzed (Participants) | 16 | 16
  Month 6 | 15.3 (4.9) | 34.3 (7.9)

16. Secondary Outcome: Pain Stages of Change Questionnaire (PSOCQ) Action Scale Score
Description: The Pain Stages of Change Questionnaire, Adolescent and Parent Report is a 30-item measure designed to evaluate parent and adolescent perceptions of readiness to adopt a self-management approach to pain. Responses are given on a 5-point scale where 1 = strongly disagree and 5 = strongly agree. Average scores are obtained for categories of Pre-contemplation (believing pain management is solely the responsibility of medical professionals), Contemplation (considering using self-management for pain), Action (starts taking ownership of pain control and self-management of pain), and Maintenance (continuous development and self-management of chronic pain); the category with the highest score indicates where the youth participant is in terms of stages of change related to pain management. For this outcome measure, the average scores for the Action scale are reported. Total scores for the Action scale range from 1 to 5 and higher scores indicate increased readiness to self-manage pain.
Time Frame: Baseline, Immediately Post-Treatment, Month 3, Month 6
Population: The analysis population includes participants remaining in the study at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Back2Life Program for Youth | Back2Life for Parents or Caregivers
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 3.7 (0.58) | 3.9 (0.45)
  Immediately Post-Treatment: number analyzed (Participants) | 16 | 16
  Immediately Post-Treatment | 3.9 (0.69) | 4.3 (0.44)
  Month 3: number analyzed (Participants) | 16 | 16
  Month 3 | 4.0 (0.45) | 3.9 (0.42)
  Month 6: number analyzed (Participants) | 16 | 16
  Month 6 | 4.2 (0.64) | 3.8 (0.98)

17. Secondary Outcome: Interleukin -1β (IL-1β) Concentration
Description: Plasma concentration of the inflammatory biomarker IL-1β is assessed among youth participants who opted for blood sample collection. IL-1β increases in response to inflammation, pain, and autoimmune diseases.
Time Frame: Baseline, Month 3, Month 6
Population: This analysis includes youth participants who provided an analyzable blood sample for the indicated time point. Collection of biomarkers was an optional study activity for participants, requiring separate consent. A total of 4 participants contributed at least one sample during the course of the study. Not all collected samples could be analyzed due to laboratory issues, such as insufficient sample volume.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Back2Life Program for Youth
Number analyzed (Participants) | 4
picograms per milliliter (pg/mL)
  Baseline: number analyzed (Participants) | 3
  Baseline | 1.25 (1.21)
  Month 3: number analyzed (Participants) | 1
  Month 3 | 1.15 (0)
  Month 6: number analyzed (Participants) | 2
  Month 6 | 0.95 (0.88)

18. Secondary Outcome: IInterleukin 6 (IL-6) Concentration
Description: Plasma concentration of the inflammatory biomarker IL-6 is assessed among youth participants who opted for blood sample collection. IL-6 is increased during injury or illness.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Back2Life Program for Youth
Number analyzed (Participants) | 4
pg/mL
  Baseline: number analyzed (Participants) | 3
  Baseline | 1.88 (2.31)
  Month 3: number analyzed (Participants) | 1
  Month 3 | 2.24 (0)
  Month 6: number analyzed (Participants) | 2
  Month 6 | 1.91 (1.80)

19. Secondary Outcome: Interleukin 8 (IL-8) Concentration
Description: Plasma concentration of the inflammatory biomarker IL-8 is assessed among youth participants who opted for blood sample collection. IL-8 is produced during the presence of inflammation.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Back2Life Program for Youth
Number analyzed (Participants) | 4
pg/mL
  Baseline: number analyzed (Participants) | 3
  Baseline | 10.28 (8.26)
  Month 3: number analyzed (Participants) | 1
  Month 3 | 27.70 (0)
  Month 6: number analyzed (Participants) | 2
  Month 6 | 14.28 (14.32)

20. Secondary Outcome: Tumor Necrosis Factor - Alpha (TNF-α) Concentration
Description: Plasma concentration of the inflammatory biomarker TNF-α is assessed among youth participants who opted for blood sample collection. TNF-α is a pro-inflammatory cytokine that regulates the inflammatory response and it is elevated during illness or injury.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Back2Life Program for Youth
Number analyzed (Participants) | 4
pg/mL
  Baseline: number analyzed (Participants) | 3
  Baseline | 2.05 (2.38)
  Month 3: number analyzed (Participants) | 1
  Month 3 | 2.57 (0)
  Month 6: number analyzed (Participants) | 2
  Month 6 | 2.04 (1.93)

21. Secondary Outcome: C-Reactive Protein (CRP) Concentration
Description: Plasma concentration of the inflammatory biomarker CRP is assessed among youth participants who opted for blood sample collection. CRP increases in response to bodily inflammation.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Back2Life Program for Youth
Number analyzed (Participants) | 4
nanograms per milliliter (ng/mL)
  Baseline: number analyzed (Participants) | 3
  Baseline | 1710.74 (746.33)
  Month 3: number analyzed (Participants) | 1
  Month 3 | 4795.63 (0)
  Month 6: number analyzed (Participants) | 2
  Month 6 | 5206.06 (3271.69)

22. Secondary Outcome: Brain-Derived Neurotrophic Factor (BDNF) Concentration
Description: Plasma concentration of the inflammatory biomarker BDNF is assessed among youth participants who opted for blood sample collection. BDNF expression is reduced when high bodily inflammation is present.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Back2Life Program for Youth
Number analyzed (Participants) | 4
pg/mL
  Baseline: number analyzed (Participants) | 3
  Baseline | 4052.33 (1445.30)
  Month 3: number analyzed (Participants) | 1
  Month 3 | 3823.00 (0)
  Month 6: number analyzed (Participants) | 2
  Month 6 | 4867.50 (1853.33)

23. Secondary Outcome: Interferon Gamma (IFN-y) Concentration
Description: Plasma concentration of the inflammatory biomarker IFN-y is assessed among youth participants who opted for blood sample collection. IFN-y is involved with regulating immune and inflammatory responses. IFN-y concentration is elevated during illness.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Back2Life Program for Youth
Number analyzed (Participants) | 4
pg/mL
  Baseline: number analyzed (Participants) | 3
  Baseline | 19.26 (17.99)
  Month 3: number analyzed (Participants) | 1
  Month 3 | 20 (0)
  Month 6: number analyzed (Participants) | 2
  Month 6 | 19.70 (10.04)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time of consent and continued through the Month 6 assessment.
Arm/Group | Back2Life Program for Youth | Back2Life for Parents or Caregivers
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT04602728/Prot_SAP_001.pdf
  • Informed Consent Form (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT04602728/ICF_000.pdf